CLINICAL TRIAL: NCT00564837
Title: Comparison of Home Vs. Physiotherapy-Supervised Rehabilitation Programs Following Reconstruction of the Anterior Cruciate Ligament (ACL)
Brief Title: Home Vs. Physiotherapy Supervised Rehabilitation After ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Calgary Health Region (Other); Olympic Oval Endowment Fund (Unknown); AirCast LLC (Industry); Fitter International Inc. (Industry)
Responsible Party: Nicholas Mohtadi, University of Calgary Sport Medicine Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10339
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: ACL Reconstruction
Keywords: Anterior cruciate ligament; Reconstruction; Rehabilitation; Home-based

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home-based (Experimental): Home-based post-operative rehabilitation program with 4 scheduled physiotherapy sessions over the first 3 post-op months
  Interventions: Procedure: Home-based rehabilitation program
- Physiotherapy supervised (Active Comparator): Physiotherapy-supervised rehabilitation program including 17 scheduled physiotherapy sessions in the first 3 post-op months
  Interventions: Procedure: Physiotherapy-supervised rehabilitation program

INTERVENTIONS:
Procedure: Home-based rehabilitation program — Home-based rehabilitation program that includes 4 physiotherapy sessions in the first 3 post-op months
  Arms: Home-based
Procedure: Physiotherapy-supervised rehabilitation program — Physiotherapy-supervised rehabilitation program that includes 17 scheduled physiotherapy sessions in the first 3 post-op months
  Arms: Physiotherapy supervised

SUMMARY:
This study was designed to determine whether or not there were any differences in knee range of motion, both statically and during gait, sagittal plane knee laxity, and quadriceps and hamstrings strength in patients three months post-ACL reconstruction with a bone-patellar tendon-bone autograft based on their performance of a primarily home based rehabilitation program or a standard physiotherapy-supervised program.

ELIGIBILITY:
Inclusion Criteria:

1. 16 years of age or older
2. Surgery at least 6 weeks after injury to allow for a return of full range of motion, minimize swelling, and offset strength deficits due to pain/swelling14,28
3. ACL reconstruction with a bone-patellar tendon-bone autograft

Exclusion Criteria:

1. Previous or concomitant reconstruction of any knee ligament to either knee
2. Ongoing knee abnormality unrelated to the ACL injury (eg, evidence of changes on radiographs consistent with osteoarthritis)
3. Professional athletes or workers' compensation patients
4. Complications during surgery (eg, inadequate graft fixation requiring protocol modification)
5. Patients without access to local physical therapy services

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 1999-09; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Active assisted knee flexion and passive knee extension range of motion | pre-op, 6 & 12 weeks post-op

SECONDARY OUTCOMES:
Knee flexion and extension range of motion during gait | pre-op, 6 & 12 wks post-op
Sagittal plane laxity of the knee | pre-op, 6 & 12 wks post-op
Isokinetic quadriceps and hamstrings strength | pre-op and 12wks post-op

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas G. Mohtadi, MD, MSc, Principal Investigator — University of Calgary Sport Medicine Centre
Locations (1):
- University of Calgary Sport Medicine Centre, Calgary, Alberta, Canada

REFERENCES:
- [Result] Grant JA, Mohtadi NG, Maitland ME, Zernicke RF. Comparison of home versus physical therapy-supervised rehabilitation programs after anterior cruciate ligament reconstruction: a randomized clinical trial. Am J Sports Med. 2005 Sep;33(9):1288-97. doi: 10.1177/0363546504273051. Epub 2005 Jul 7. PMID 16002493